CLINICAL TRIAL: NCT00665509
Title: Immunogenicity, Reactogenicity and Safety of the Trivalent Influenza Subunit Vaccine Influvac® for the Season 2008/2009. An Open-Label, Baseline-Controlled Multi-Center Study in Two Groups: Adult Subjects and Elderly Subjects
Brief Title: Annual Study to Investigate Inactivated Subunit Influenza Vaccine Due to New Virus Strains for the 08/09 Season.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Biologicals (Industry)
Responsible Party: Maaike Cronenberg, Solvay Pharmaceuticals
Organization: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S201.3.127; 2008-001038-28
Record Dates: First submitted 2008-04-10; First posted 2008-04-24 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; CHMP criteria
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Trivalent influenza subunit vaccine Influvac

INTERVENTIONS:
Biological: Trivalent influenza subunit vaccine Influvac — 3x 15mcg HA per 0.5 ml, trivalent one injection at Day 1

SUMMARY:
Influenza (flu) viruses change continuously, therefore also the parts of viruses used in influenza vaccines can vary from year to year. In Europe, manufacturers/marketing holders of these vaccines are required to be involved in ongoing clinical trials and to present the results to the competent authorities each year. The current study is a phase IIIa clinical trial with a commercially available vaccine (Influvac®) supplied in pre filled syringes. It is part of the ongoing clinical trial program for Influvac® and will be done to assess the immunogenicity and safety and tolerability of next season's trivalent influenza subunit vaccine in two groups of healthy subjects: subjects aged >= 18 and <= 60 years and subjects >= 61 years of age (elderly).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent and able to adhere to all protocol required study procedures.
* Men and women aged ≥ 18 and ≤ 60 years or ≥ 61 years of age at the day of study vaccination.
* Being in good health as judged by medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

* Known to be allergic to eggs, chicken protein, gentamicin or any other constituent of the vaccine.
* A serious adverse reaction after a previous (influenza) vaccination. Presence of any significant condition that may prohibit inclusion as determined by the investigator.
* Having received vaccination against influenza within the previous six months before study vaccination or planned vaccination during the study period.
* A history of Guillain-Barré syndrome or active neurological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity (HI-titers after 2 and 3 weeks), reactogenicity and inconvenience of Influvac® 2008/2009 | 2 and 3 weeks

SECONDARY OUTCOMES:
HI derived parameters: seroprotection, seroconversion and mean fold increase (CHMP) | 2 and 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (2):
- Site 1, Tessenderlo, Belgium
- Site 2, Hamburg, Germany